CLINICAL TRIAL: NCT00884286
Title: A Phase II Multicenter, Open-Label, Clinical And Pharmacokinetic Study of Aplidin® As A 1-Hour Weekly IV Infusion, in Patients With Relapsed Or Refractory Aggressive Non-Hodgkin's Lymphoma
Brief Title: Multicenter Trial to Treat Patients With Relapsed/Refractory Aggressive Non Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APL-B-013-02
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2011-02

CONDITIONS: Leukemia; Lymphoma
Keywords: Aplidin; Aggressive Non Hodgkin Lymphoma; Leukemia-Lymphoma, Adult T-Cell and B-cell
MeSH Terms: conditions — Leukemia; Lymphoma | interventions — plitidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm One (Experimental): Aplidin® given as a 1-hour weekly IV infusion
  Interventions: Drug: Aplidin®

INTERVENTIONS:
Drug: Aplidin® — Aplidin® will be administered at a starting dose of 3.2 mg/m2, as a 1-hour intravenous infusion, on days 1, 8 and 15, every 28 days cycle.
  Other Names: plitidepsin

SUMMARY:
This is a multicenter study to assess the anti-tumour activity,to investigate the safety profile and to obtain additional pharmacokinetic information for Aplidin® given as 1-hour weekly IV infusion in patients with aggressive non-Hodgkin's Lymphoma.

DETAILED DESCRIPTION:
A Phase II Multicenter,Open-Label, Clinical And Pharmacokinetic Study Of Aplidin® As A 1-Hour Weekly IV Infusion, In Patients With Relapsed Or Refractory aggressive non-Hodgkin's Lymphoma.

Primary

• To assess the anti-tumour activity of Aplidin® given as a 1-hour weekly IV infusion, in patients with aggressive non-Hodgkin's Lymphoma, relapsing or refractory to a prior therapy.

Secondary

* To further investigate the safety profile of Aplidin® given as 1-hour weekly IV infusion in this patient population.
* To obtain additional pharmacokinetic information for Aplidin® given as 1-hour weekly IV infusion in patients with aggressive non-Hodgkin's Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Histologically confirmed aggressive lymphomas,
* Patient requires treatment because NHL relapses
* Measurable disease
* Recovery from any non-hematological toxicity derived from previous treatments. The presence of alopecia and NCI-CTC grade < 2 symptomatic peripheral neuropathy is allowed.
* Age > 18 years.
* Performance status (ECOG) < 2
* Adequate renal, hepatic, and bone marrow function (assessed < 14 days before inclusion in the study)
* Left ventricular ejection fraction within normal limits.

Exclusion Criteria:

* Prior therapy with Aplidin®.
* Concomitant therapy with any anti-lymphoproliferative agent
* Acute lymphoblastic leukemia.
* CNS lymphoma.
* HIV-associated lymphoma.
* Prior gene therapy with viral vectors.
* More than three previous lines of systemic biological agents or chemotherapies. Wash-out periods since the end of the precedent therapy less than:

  * 6 weeks for nitroso-urea or high dose chemotherapy
  * 3 weeks for other chemotherapies or biological agents
  * 4 weeks for radiation or radionuclide therapy (6 weeks in case of prior extensive external beam radiation (more than 25% of bone marrow distribution).
  * 4 weeks for major prior surgery
  * 30 days for any investigational product
  * 4 weeks for immunosuppressive therapy after allogeneic hematopoietic stem cell transplantation.
* Pregnant or lactating women.
* Men and women of reproductive potential who are not using effective contraceptive methods
* History of another neoplastic disease. Exceptions: Non-melanoma skin cancer,cCarcinoma in situ of any site,any other cancer curatively treated and no evidence of disease for at least 10 years.
* Known cerebral or leptomeningeal involvement.
* Other relevant diseases or adverse clinical conditions
* Treatment with any investigational product in the 30 days period before inclusion in the study.
* Known hypersensitivity to Aplidin®, mannitol, cremophor EL, or ethanol
* Limitation of the patient's ability to comply with the treatment or follow-up protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2004-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Ribrag, MD, Principal Investigator — Institut Gustave Roussy, France
Locations (12):
- France (3):
  - Centre Hospitalier Lyon Sud, Lyon
  - Hôpital Saint- Louis, Paris
  - Institut Gustave Roussy, Villejuif
- Italy (3):
  - Istituto di ematologia e oncologia medica "L. e. A. Seragnoli", Bologna
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Ospedaliero Universitaria de Modena, Modena
- Instituto Nacional de Enfermedades Neoplásicas (INEN), Surquillo, Lima region, Peru
- Hospital Español Auxilio Mutuo de Puerto Rico Inc., San Juan, Puerto Rico
- Spain (3):
  - Hospital Clinico de Barcelona, Barcelona
  - Hospital Morales Meseguer, Murcia
  - Hospital Universitario de Salamanca, Salamanca
- Istituto Oncologico della Svizzera Italiana - Ospedale San Giovanni, Bellinzona, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ribrag V, Caballero D, Ferme C, Zucca E, Arranz R, Briones J, Gisselbrecht C, Salles G, Gianni AM, Gomez H, Kahatt C, Corrado C, Szyldergemajn S, Extremera S, de Miguel B, Cullell-Young M, Cavalli F. Multicenter phase II study of plitidepsin in patients with relapsed/refractory non-Hodgkin's lymphoma. Haematologica. 2013 Mar;98(3):357-63. doi: 10.3324/haematol.2012.069757. Epub 2012 Oct 12. PMID 23065525

RESULTS

PARTICIPANT FLOW:
Groups:
- Aplidin® (Cohort Non-cutaneous PTCL); Aplidin®(Other Lymphoma): Aplidin® given as a 1-hour weekly IV infusion
  Aplidin®: Aplidin® will be administered at a starting dose of 3.2 mg/m2, as a 1-hour intravenous infusion, on days 1, 8 and 15, every 28 days cycle.
Period: Overall Study
Arm/Group | Aplidin® (Cohort Non-cutaneous PTCL) | Aplidin®(Other Lymphoma)
Started | 34 | 33
Completed | 2 | 0
Not Completed | 32 | 33
Not completed — Progressive disease | 21 | 28
Not completed — Toxicity | 4 | 1
Not completed — Death | 2 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Septic shock | 1 | 0
Not completed — Thrombus in right auricle | 1 | 0
Not completed — Not treated | 2 | 1
Not completed — Comprised lung carcinoma | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Aplidin® (Cohort Non-cutaneous); Aplidin® (Cohort Other Lymphoma): Aplidin® given as a 1-hour weekly IV infusion
  Aplidin®: Aplidin® will be administered at a starting dose of 3.2 mg/m2, as a 1-hour intravenous infusion, on days 1, 8 and 15, every 28 days cycle.
- Total: Total of all reporting groups
Arm/Group | Aplidin® (Cohort Non-cutaneous) | Aplidin® (Cohort Other Lymphoma) | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Customized [Count of Participants; unit: Participants] — A 17 year-old patient was included and it was considered by the Sponsor as a non-clinically relevant protocol deviation.
  Participants
    17 years | 0 | 1 | 1
    Between 18 and 49 years | 14 | 3 | 17
    Between 50 and 69 years | 14 | 19 | 33
    >= 70 years | 6 | 10 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 22 | 46
  Male | 10 | 11 | 21
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 3 | 0 | 3
  France | 20 | 23 | 43
  Switzerland | 2 | 1 | 3
  Peru | 2 | 0 | 2
  Spain | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: The primary objective of the study was the exploration of the efficacy of plitidepsin when given as a weekly 1-hour infusion on Days 1, 8 and 15 in 4-week cycles to patients with relapsed or refractory aggressive non-Hodgkin's Lymphoma.
  The primary efficacy endpoint was the Objective Response Rate, defined as the combined rate of Complete Response (CR), Unconfirmed Complete Response (CRu) and Partial Response (PR) following the definition of response according to the International Working Group (IWG) criteria for Non-Hodgkin's Lymphoma (NHL).
Time Frame: All patients were followed up to progressive disease, start of a new anti-cancer therapy, death or one year after the last treatment visit of the last patient, whichever occured first
Population: The efficacy and safety analyses were to be performed separately for the subset of treated patients with non-cutaneous Peripheral T-cell Lymphoma (PTCL), and for the subset of treated patients with other lymphomas.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm One
Number analyzed (Participants) | 67
Participants
  Non-cutaneous PTCL: number analyzed (Participants) | 34
  Non-cutaneous PTCL: Complete response | 2
  Non-cutaneous PTCL: Partial response | 4
  Non-cutaneous PTCL: Stable Disease | 6
  Non-cutaneous PTCL: Progressive disease | 17
  Non-cutaneous PTCL: Not evaluable | 5
  Other lymphomas: number analyzed (Participants) | 33
  Other lymphomas: Complete response | 0
  Other lymphomas: Partial response | 0
  Other lymphomas: Stable Disease | 6
  Other lymphomas: Progressive disease | 24
  Other lymphomas: Not evaluable | 3

2. Secondary Outcome: Time to Response Onset
Description: Time to response onset was defined as the time from the first day of plitidepsin treatment to the first documentation of response.
Time Frame: as for outcome 1
Population: The efficacy and safety analyses were to be performed separately for the subset of treated patients with non-cutaneous PTCL, and for the subset of treated patients with other lymphomas.
  Six responders belong to the Non-cutaneous PTCL cohort
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Arm One (Non-cutaneous PTCL Cohort): Aplidin® given as a 1-hour weekly IV infusion
  Aplidin®: Aplidin® will be administered at a starting dose of 3.2 mg/m2, as a 1-hour intravenous infusion, on days 1, 8 and 15, every 28 days cycle.
Arm/Group | Arm One (Non-cutaneous PTCL Cohort)
Number analyzed (Participants) | 6
weeks | 7.5 [6.9 to 7.9]

3. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from the first documented objective response (CR, CRu or PR) to disease progression or death. Patients who had not progressed or died were to have their duration censored at the date of their last disease assessment.
Time Frame: as for outcome 1
Population: The efficacy and safety analyses were to be performed separately for the subset of treated patients with non-cutaneous PTCL, and for the subset of treated patients with other lymphomas.
  The six responders belong to the Non-cutaneous PTCL cohort.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm One (Non-cutaneous PTCL Cohort)
Number analyzed (Participants) | 6
months | 2.2 [0 to 27.9]

4. Secondary Outcome: Time to Progression
Description: Time to progression (TTP) was to be calculated from the first day of plitidepsin treatment to the date of disease progression.
Time Frame: as for outcome 1
Population: The efficacy and safety analyses were to be performed separately for the subset of treated patients with non-cutaneous PTCL, and for the subset of treated patients with other lymphomas.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm One
Number analyzed (Participants) | 59
months
  Non-cutaneous PTCL: number analyzed (Participants) | 29
  Non-cutaneous PTCL | 1.6 [1.1 to 3.0]
  Other lymphomas: number analyzed (Participants) | 30
  Other lymphomas | 1.3 [0.8 to 1.6]

5. Secondary Outcome: Time to Subsequent Chemotherapy
Description: Time to subsequent therapy was to be calculated from the first infusion of the study drug to the start date of the subsequent therapy. Patients without subsequent therapy were to be censored at their last reported date.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm One (Subset of Treated Patients With Other Lymphomas): Aplidin® given as a 1-hour weekly IV infusion
  Aplidin®: Aplidin® will be administered at a starting dose of 3.2 mg/m2, as a 1-hour intravenous infusion, on days 1, 8 and 15, every 28 days cycle.
Arm/Group | Arm One (Non-cutaneous PTCL Cohort) | Arm One (Subset of Treated Patients With Other Lymphomas)
Number analyzed (Participants) | 32 | 32
months | 3.8 [2.3 to 5.6] | 1.9 [1.4 to 2.6]

6. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was to be calculated from the date of registration to the date of first objective disease progression or death from any cause. Patients who were lost to follow-up without documentation of progression were to be censored at the last date they were assessed and found progression-free.
  A patient receiving a new treatment in the absence of documented progression was to be considered as progressing at the time of re-treatment.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm One
Number analyzed (Participants) | 59
months
  Non-cutaneous PTCL: number analyzed (Participants) | 29
  Non-cutaneous PTCL | 1.6 [1.1 to 2.7]
  Other lymphomas: number analyzed (Participants) | 30
  Other lymphomas | 1.3 [0.8 to 1.6]

7. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was to be calculated from the date of registration to the date of death from any cause. Patients with no documented death were to be censored at the last date they were known to be alive.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm One
Number analyzed (Participants) | 59
months
  Non-cutaneous PTCL: number analyzed (Participants) | 29
  Non-cutaneous PTCL | 10.2 [4.4 to 24.3]
  Other lymphomas: number analyzed (Participants) | 30
  Other lymphomas | 4.5 [2.7 to 6.4]

ADVERSE EVENTS:
Description: Only 64 out of 67 included patients were treated, therefore, 64 patients were considered as participant at risk.
Groups:
- Aplidin® (Cohort Other Lymphomas): Aplidin® given as a 1-hour weekly IV infusion
  Aplidin®: Aplidin® will be administered at a starting dose of 3.2 mg/m2, as a 1-hour intravenous infusion, on days 1, 8 and 15, every 28 days cycle.
Arm/Group | Aplidin® (Cohort Non-cutaneous PTCL) | Aplidin® (Cohort Other Lymphomas)
All-Cause Mortality (participants affected / at risk) | 10/32 | 10/32
Serious Adverse Events (participants affected / at risk) | 13/32 | 11/32
Other Adverse Events (participants affected / at risk) | 31/32 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aplidin® (Cohort Non-cutaneous PTCL) (N=32) | Aplidin® (Cohort Other Lymphomas) (N=32)
Abdominal pain NOS (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage NOS (Gastrointestinal disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Diarrhea NOS (Gastrointestinal disorders) | 0 | 1
Atrial thrombosis (Cardiac disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
Condition aggravated (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 3
Rigors (General disorders) | 1 | 0
Disease progression NOS (General disorders) | 0 | 1
Injection site reaction NOS (General disorders) | 1 | 0
Cardiac troponin I increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Anemia NOS (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Guillain-Barré syndrome (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysponea NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Obstructive airways disorder NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension NOS (Vascular disorders) | 1 | 0
Enteritis necroticans (Infections and infestations) | 1 | 0
Gastroenteritis NOS (Infections and infestations) | 1 | 0
Pneumonia NOS (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 2 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aplidin® (Cohort Non-cutaneous PTCL) (N=32) | Aplidin® (Cohort Other Lymphomas) (N=32)
Anaemia NOS (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Leukopenia NOS (Blood and lymphatic system disorders) | 2 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Arrhythmia NOS (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Bradycardia NOS (Cardiac disorders) | 0 | 1
Cardiac flutter (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Supraventricular arrhythmia NOS (Cardiac disorders) | 1 | 0
Tachycardia NOS (Cardiac disorders) | 4 | 1
Ventricular arrhythmia NOS (Cardiac disorders) | 0 | 1
Ventricular hypokinesia (Cardiac disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Acquired hypothyroidism (Endocrine disorders) | 1 | 0
Cushingoid (Endocrine disorders) | 1 | 0
Eye inflammation NOS (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Eyelid oedema (Eye disorders) | 1 | 0
Ophthalmoplegia NOS (Eye disorders) | 1 | 0
Uveitis NOS (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Visual disturbance NOS (Eye disorders) | 1 | 0
Abdominal pain NOS (Gastrointestinal disorders) | 6 | 4
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3
Aptyalism (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 6
Diarrhoea NOS (Gastrointestinal disorders) | 10 | 7
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Dysphagia (Gastrointestinal disorders) | 2 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction NOS (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 11 | 13
Oesophageal pain (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Rectal tenesmus (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting NOS (General disorders) | 5 | 5
Chest pain (General disorders) | 0 | 2
Condition aggravated (General disorders) | 1 | 0
Fatigue (General disorders) | 20 | 19
General physical health deterioration (General disorders) | 1 | 0
Inflammation NOS (General disorders) | 1 | 0
Inflammation localised (General disorders) | 1 | 0
Oedema NOS (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 5 | 13
Pain NOS (General disorders) | 1 | 1
Pyrexia (General disorders) | 16 | 4
Rigors (General disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 1
Abscess NOS (Infections and infestations) | 1 | 0
Bacterial infection NOS (Infections and infestations) | 0 | 1
Candidal infection NOS (Infections and infestations) | 1 | 1
Clostridial infection NOS (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Eye infection NOS (Infections and infestations) | 0 | 1
Fungal infection NOS (Infections and infestations) | 0 | 1
Infection NOS (Infections and infestations) | 1 | 0
Infectious mononucleosis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Pneumocystis carinii infection (Infections and infestations) | 0 | 1
Pseudomonas infection NOS (Infections and infestations) | 0 | 1
Sinusitis NOS (Infections and infestations) | 2 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Tonsillitis NOS (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood alkaline phosphatase NOS increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 2
Blood urine present (Investigations) | 1 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 2
Weight decreased (Investigations) | 7 | 3
Weight increased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 9 | 5
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia NOS (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle cramps (Musculoskeletal and connective tissue disorders) | 3 | 4
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 3 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 11
Myopathy toxic (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in limb (Musculoskeletal and connective tissue disorders) | 1 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 9
Aphonia (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1
Dysphonia (Nervous system disorders) | 0 | 1
Headache NOS (Nervous system disorders) | 2 | 1
Hyperaesthesia (Nervous system disorders) | 1 | 0
Hyporeflexia (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 3 | 4
Peripheral neuropathy NOS (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Vasovagal attack (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 2
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Libido decreased (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Haemoglobinuria (Renal and urinary disorders) | 0 | 1
Incontinence NOS (Renal and urinary disorders) | 0 | 1
Polyuria (Renal and urinary disorders) | 1 | 0
Renal failure NOS (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Breath sounds decreased (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung crepitation (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lung disorder NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural disorder NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sputum abnormal NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 4 | 2
Erythrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Pigmentation disorder NOS (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus NOS (Skin and subcutaneous tissue disorders) | 6 | 2
Rash NOS (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin eruption (Skin and subcutaneous tissue disorders) | 1 | 1
Skin lesion NOS (Skin and subcutaneous tissue disorders) | 1 | 0
Sweating increased (Skin and subcutaneous tissue disorders) | 5 | 1
Deep venous thrombosis NOS (Vascular disorders) | 0 | 1
Hypotension NOS (Vascular disorders) | 2 | 0
Lymphangitis (Vascular disorders) | 0 | 1
Lymphoedema NOS (Vascular disorders) | 1 | 0
Pallor (Vascular disorders) | 0 | 6
Peripheral coldness (Vascular disorders) | 1 | 0
Peripheral revascularisation (Vascular disorders) | 1 | 0
Phlebitis NOS (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days